CLINICAL TRIAL: NCT04485819
Title: Achieving Better Clinical Outcomes With Blastocyt Transfer in Poor Responders: a Prospective Study
Brief Title: Optimal Embryonic Stage for Transfer in Poor Responders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Other Study IDs: MH0003
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Poor Response to Ovulation Induction; Infertility, Female
Keywords: Poor responders; Embryo transfer; Cancellation rate; Implantation rate; Live birth rate
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cleavage stage transfer: Poor responders who transfer their embryos in cleavage stage on day 3
  Interventions: Other: Cleavage stage transfer
- Blast stage transfer: Poor responders who transfer their embryos on blast stage on day 5/6
  Interventions: Other: Blast stage transfer

INTERVENTIONS:
Other: Cleavage stage transfer — transferring embryos through ICSI procedures for poor responders on cleavage stage of embryonic development.
  Groups: Cleavage stage transfer
Other: Blast stage transfer — transferring embryos through ICSI procedures for poor responders on blast stage of embryonic development.
  Groups: Blast stage transfer

SUMMARY:
A Prospective cohort study including couples with poor responder females who undergoing ICSI

DETAILED DESCRIPTION:
Purpose:

To determine the optimal embryonic stage for transfer in poor responders.

Method:

Patients were divided into day 3 transfer group and day 5 transfer group. All cases had the same stimulation protocol and planning to do fresh embryo transfer. Assessments will be at Day 1, Day 3 and Day 5/6 according to Gardner's criteria 1999. Embryological and clinical data were recorded and then analyzed using SPSS (version 23) statistical software.

ELIGIBILITY:
Inclusion Criteria:

* poor responders females with AMH≤ 1.2ng and have ≤ 5 mature oocytes
* couples whose planning to do fresh transfer
* male partners have normal semen parameters according to WHO 2010.

Exclusion Criteria:

* sperm or oocyte donation
* gestational carriers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — poor responders females with AMH≤ 1.2ng and have ≤ 5 mature oocytes
Study Population: Poor responders undergoing ICSI procedures at Ganin fertility center in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | delivery of healthy neonate after 37 weeks of pregnancy
  percentage of cycles started with the intent of egg retrieval that led to a live birth.
Implantation rate | 6 weeks of pregnancy
  Percentage of the implanted embryos number for each group / number of transferred embryos.

SECONDARY OUTCOMES:
Clinical pregnancy rate | after 6 weeks of embryonic transfer
  Percentage of pregnant cases with fetal heart / transferred cases for each group
Cancellation rate | 5:6 days of ICSI
  percentage of blast transfer cases who did not achieve blast stage (cancelled cases) / total number of blast stage cases
Fertilization rate | 16:19 hours after intracytoplasmic injection(ICSI)
  Percentage of fertilized oocyte (appearance of two pronuclei) / Number of injected oocytes
Cleavage rate | 72 hours after ICSI
  Percentage of cleaved embryos / Number of fertilized oocytes
High quality day 3 embryos | 72 hours after ICSI
  High quality D3 embryos according to Gardner's criteria / total cleaved embryos
Blast rate | 5:6 days of ICSI
  Percentage of total blastocysts / Total cleaved embryos
High quality blast rate | 5:6 days of ICSI
  Morphological grading of trophectoderm and Inner cell mass using Gardner's criteria 1999, from grade A and B ( A is the highest quality). Total high grade embryos/ total blast embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Manar Hozyen, MSc., Principal Investigator — Ganin Fertility Center; Amira Hassan, BSc., Principal Investigator — Ganin Fertility Center; Hanaa Elkhader, BSc., Principal Investigator — Ganin Fertility Center; Hosam Zaki, Study Chair — Ganin Fertility Center
Locations (1):
- Ganin fertility center, Cairo, Egypt